CLINICAL TRIAL: NCT02965716
Title: A Phase II Study of Combining Talimogene Laherparepvec (T-VEC) (NSC-785349) and MK-3475 (Pembrolizumab) (NSC-776864) in Patients With Advanced Melanoma Who Have Progressed on Anti-PD1/L1 Based Therapy
Brief Title: Talimogene Laherparepvec and Pembrolizumab in Treating Patients With Stage III-IV Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2016-01698; NCI-2016-01698 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1607; S1607 (Other: SWOG); S1607 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2016-11-16; First posted 2016-11-17 (Estimated); Results first posted 2024-08-27 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Advanced Melanoma; Recurrent Melanoma; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (talimogene laherparepvec, pembrolizumab) (Experimental): Patients receive talimogene laherparepvec IL and pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Biological: Talimogene Laherparepvec

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Biological: Talimogene Laherparepvec — Given IL
  Other Names: ICP34.5-, ICP47-deleted Herpes Simplex Virus 1 (HSV-1) Incorporating the Human GM-CSF Gene; Imlygic; JS1 34.5-hGMCSF 47- pA-; T-VEC

SUMMARY:
This phase II trial studies how well talimogene laherparepvec and pembrolizumab work in treating patients with stage III-IV melanoma. Biological therapies, such as talimogene laherparepvec, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop tumor cells from growing. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving talimogene laherparepvec and pembrolizumab may work better in treating patients with melanoma by shrinking the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the objective response rate (confirmed complete and partial responses) of treatment with talimogene laherparepvec (T-VEC) in combination with pembrolizumab (MK-3475) following progression on prior anti-PD-1 or anti-PD-L1 therapy alone or in combination with other agents different from talimogene laherparepvec (T-VEC).

SECONDARY OBJECTIVES:

I. To estimate the durable response rate. II. To estimate the objective response rate (ORR) defined as confirmed and unconfirmed, complete and partial responses in the injected lesions.

III. To estimate the ORR in the non-visceral, non-injected lesions. IV. To estimate the ORR in the visceral lesions (Cohort A). V. To estimate the median progression-free survival (PFS). VI. To estimate the median overall survival (OS). VII. To evaluate the toxicity of the regimen.

TRANSLATIONAL OBJECTIVES:

I. To evaluate whether adding talimogene laherparepvec (T-VEC) to PD1 blockade can increase T-cell infiltration into tumors and whether change in T-cell infiltration is associated with response.

II. To evaluate whether adding talimogene laherparepvec (T-VEC) to PD1 blockade can increase T-cell receptor (TCR) clonality in tumors and in peripheral blood and whether increased TCR clonality is associated with response.

III. To evaluate whether intra-tumoral injection of talimogene laherparepvec (T-VEC) can improve the tumor immune microenvironment.

IV. To evaluate whether tumor mutational load, mutations in the IFN pathway, and circulating tumor deoxyribonucleic acid (DNA) profile are is associated with response to talimogene laherparepvec (T-VEC) plus pembrolizumab (MK-3475) therapy in the anti-PD1/L1 therapy refractory melanoma patients.

OUTLINE:

Patients receive talimogene laherparepvec intralesionally (IL) and pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for up to 1 year and then annually for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed stage IV or unresectable stage III melanoma; patients must not have disease that is suitable for local therapy, administered with curative intent
* Patients must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; contrast-enhanced computed tomography (CT) scans of the chest, abdomen and pelvis are required; a whole body positron emission tomography (PET)/CT scan with diagnostic quality images and intravenous iodinated contrast may be used in lieu of a contrast enhanced CT of the chest, abdomen and pelvis; imaging of the head and neck, or the limbs is required only if the patient has a lesion(s) in these areas; contrast may be omitted if the treating investigator believes that exposure to contrast poses an excessive risk to the patient; if skin lesions are being followed as measurable disease, photograph with a ruler included and physician's measurements, must be kept in the patients chart as source documentation; all measurable lesions must be assessed within 28 days prior to registration; tests to assess non-measurable disease must be performed within 42 days prior to registration.; all disease must be assessed and documented on the baseline tumor assessment form (RECIST 1.1)
* Cohort A: Patients must have at least one measurable visceral lesion (per RECIST 1.1); a visceral lesion is any solid organ except for skin, lymph node, and musculoskeletal tissue; at least one of these visceral lesions must be measurable per RECIST 1.1
* Patients must, in the opinion of the treating physician, be candidates for intralesional administration into cutaneous, subcutaneous, or nodal lesions
* Patients may have brain metastases if all lesions have been treated with stereotactic radiation therapy, craniotomy, or gamma knife therapy and have not required steroids for at least 14 days prior to registration
* Patient must have had prior treatment with anti-PD-1 or anti-PD-L1 agents and have documented disease progression on these agents prior to registration; patients who have progressed after adjuvant anti-PD1/L1 agents are eligible
* Patients must be >= 18 years of age
* Patients must have Zubrod performance status =< 2
* Absolute neutrophil count (ANC) >= 1,500/mcL (within 28 days prior to registration)
* Hemoglobin >= 8 g/dL (within 28 days prior to registration)
* Platelets >= 100,000/mcL (within 28 days prior to registration)
* Albumin >= 2.5 g/dL (within 28 days prior to registration)
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN) except patients with documented Gilbert's syndrome (=< 3 x IULN is eligible) (within 28 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both =< 3 x IULN (within 28 days prior to registration)
* Patients must have lactate dehydrogenase (LDH) obtained prior to registration
* Patients must have complete physical examination and medical history obtained within 28 days prior to registration
* Patients must be offered the opportunity to submit archival tissue for translational medicine; patients must also be willing to undergo biopsies and submit tissue and blood for translational medicine; with patients consent, any remaining specimens will be banked for future use
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Exclusion Criteria:

* Cohort B: Patients must not have any visceral lesions
* Patients must not have had surgery, biologic therapy, or hormonal therapy within 14 days prior to registration; patients must not have had chemotherapy, targeted small molecule therapy, or radiation therapy within 14 days prior to registration; patients must not have had a monoclonal antibody for cancer treatment, except anti-PD1/L1 antibodies, within 28 days prior to registration

  * Patients must have recovered from all adverse events due to prior anti-cancer therapy (residual toxicity =< grade 1) prior to registration, with the exception of patients with =< grade 2 neuropathy, =< grade 2 hypothyroidism, or =< grade 2 alopecia
  * If patients received major surgery, they must have recovered adequately from toxicity and/or complications from the intervention prior to registration
* Patients must not have received prior treatment with talimogene laherparepvec (T-VEC); prior treatment with T-VEC is defined as receiving at least one injection with 1 x 10^8 plaque forming units (pfu)
* Patients must not have received any live vaccine within 30 days prior to registration; seasonal flu vaccines that do not contain live virus are permitted
* Patients must not be planning to receive other biologic therapy, radiation therapy, hormonal therapy, chemotherapy, surgery, or other therapy while on this protocol; palliative radiation therapy or surgery can be considered for symptomatic non-target lesions after discussions with the study team
* Patients must not require use of systemic corticosteroid within 14 days prior to registration or during protocol treatment; patients with preexisting severe autoimmune disease requiring systemic corticosteroids or ongoing immunosuppression are not eligible
* Patients must not have known history of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) due to contraindication of talimogene laherparepvec (T-VEC) in immune-compromised patients and that administration of talimogene laherparepvec (T-VEC) has not been tested in HIV-positive patients; the use of physiologic doses of corticosteroids may be approved after consultation with the study chair
* Patients must not have history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Patients must not have an active infection requiring systemic therapy nor a viral infection requiring intermittent treatment with an antiherpetic drug, other than intermittent topical use
* Patients must not have active herpetic skin lesions or prior complications of herpetic infection (e.g., herpetic keratitis or encephalitis) which requires intermittent or chronic treatment with an anti-herpetic drug other than intermittent topical use
* Patients must not have organ allografts
* Patients must not have an uncontrolled intercurrent illness or whose control may be jeopardized by the treatment with the study therapy, or psychiatric illness/social situations which would limit compliance with study requirements
* Patients must not have active autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other) that requires systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in the past 2 years; replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease
* Patient must not have evidence of any clinically significant immunosuppression such as the following:

  * Primary immunodeficiency state such as severe combined immunodeficiency disease;
  * Concurrent opportunistic infection;
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 2 months prior to enrollment
* Patients must not have any other malignancy that requires active treatment
* Patients must not be pregnant or nursing due to risk of fetal or nursing infant harm; women of reproductive potential must have a negative serum pregnancy test within 7 days prior to registration; women/men of reproductive potential must have agreed to use an effective contraceptive method while on study and for 120 days after last study treatment; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2026-11-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Siwen Hu-Lieskovan, Principal Investigator — SWOG Cancer Research Network
Locations (20):
- United States (20):
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Allegiance Health, Jackson, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 43 participants were enrolled to the study, 4 participants were determined to be ineligible, and 1 was not analyzable.
Groups:
- Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab): Cohort A (Visceral): Patients will take up to 4 ml of 1 million PFU/mL T-VEC intralesionally on cycle 1, and up to 4 ml of 100 million PFU/mL T-VEC intralesionally on cycles 2-36, as well as 200 mg of Pembrolizumab taken by IV over 30 minutes on cycles 1-36.
- Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab): Cohort B (Non-Visceral): Patients will take up to 4 ml of 1 million PFU/mL T-VEC intralesionally on cycle 1, and up to 4 ml of 100 million PFU/mL T-VEC intralesionally on cycles 2-36, as well as 200 mg of Pembrolizumab taken by IV over 30 minutes on cycles 1-36.
Period: Overall Study
Arm/Group | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab)
Started | 11 | 27
Completed | 0 | 3
Not Completed | 11 | 24
Not completed — Refusal Unrelated to Adverse Event | 1 | 5
Not completed — Progression/Relapse | 8 | 16
Not completed — Death | 1 | 0
Not completed — Not Protocol Specified | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab) | Total
Number analyzed (Participants) | 11 | 27 | 38
Age, Continuous [Median (Full Range); unit: years] | 61.8 [20.7 to 76.8] | 61.3 [36.1 to 93.7] | 61.55 [20.7 to 93.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 4 | 16 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 8 | 24 | 32
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 8 | 23 | 31
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 2 | 4
Performance Status [Count of Participants; unit: Participants] — Zubrod performance status scale ranges from 0 to 4, with higher scores reflecting greater disability.
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    0 | 3 | 14 | 17
    1 | 7 | 11 | 18
    2 | 1 | 2 | 3
Resistance To Prior Checkpoint Inhibitor [Count of Participants; unit: Participants] — Acquired resistance signifies that participant had responded to treatment but then progressed. Primary resistance signifies that participant had not initially responded to treatment.
  Participants
    Acquired | 3 | 3 | 6
    Primary | 8 | 24 | 32

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Number of participants with a complete response, defined as the disappearance of all target and non-target lesions, or partial response, defined as a greater than or equal to 30% decrease under baseline of the sum of appropriate diameters of all target measurable legions. ORR is measured using RECIST 1.1 guidelines.
Time Frame: Up to 5 years post registration or until death
Population: Participants who are eligible and analyzable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 11 | 27
Participants
  Complete Response | 0 | 2
  Partial Response | 0 | 5

2. Secondary Outcome: Durable Response Rate
Description: Number of participants with complete or partial response per RECIST 1.1 with no evidence of disease progression for at least 180 days from the initial documentation of CR/PR.
Time Frame: Up to 5 years post registration or until death
Population: Participants who are eligible and analyzable.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 11 | 27
participants | 0 [0 to 28] | 4 [4 to 34]

3. Secondary Outcome: Objective Response Rate (ORR) in Injected Lesions
Description: Number of participants with confirmed and unconfirmed complete and partial responses in injected lesions. A confirmed complete response (CR) is defined as 2 or more consecutive objective statuses of CR a minimum of 4 weeks apart, a confirmed partial response is defined as 2 or more consecutive objective statuses of PR or better a minimum of 4 weeks apart but no qualifying as a CR. A unconfirmed CR is defined as 1 objective status of CR but not qualifying as a CR or PR, a unconfirmed PR is defined as 1 objective status of PR but not qualifying as CR, PR, or unconfirmed CR. ORR is measured per RECIST 1.1 guidelines.
Time Frame: Up to 5 years post registration or until death
Population: Participants who are eligible and analyzable and had lesions deemed injectable at any time prior to progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 11 | 27
Participants
  Complete Response | 0 | 2
  Partial Response | 0 | 4
  Unconfirmed Complete Response | 1 | 2

4. Secondary Outcome: Objective Response Rate (ORR) in Non-Visceral, Non-Injected Lesions
Description: Number of participants with confirmed and unconfirmed complete and partial responses in non-visceral, non-injected lesions. A confirmed complete response (CR) is defined as 2 or more consecutive objective statuses of CR a minimum of 4 weeks apart, a confirmed partial response is defined as 2 or more consecutive objective statuses of PR or better a minimum of 4 weeks apart but no qualifying as a CR. A unconfirmed CR is defined as 1 objective status of CR but not qualifying as a CR or PR, a unconfirmed PR is defined as 1 objective status of PR but not qualifying as CR, PR, or unconfirmed CR. ORR is measured per RECIST 1.1 guidelines.
Time Frame: Up to 5 years post registration or until death
Population: Eligible participants who had lesions that were not injected at Cycle 1, Week 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 8 | 19
Participants
  Complete Response | 0 | 2
  Partial Response | 0 | 1
  Unconfirmed Complete Response | 0 | 1
  Unconfirmed Partial Response | 0 | 1

5. Secondary Outcome: Objective Response Rate (ORR) in Visceral Lesions (Cohort A)
Description: Number of participants with confirmed and unconfirmed complete and partial responses in visceral lesions. A confirmed complete response (CR) is defined as 2 or more consecutive objective statuses of CR a minimum of 4 weeks apart, a confirmed partial response is defined as 2 or more consecutive objective statuses of PR or better a minimum of 4 weeks apart but no qualifying as a CR. A unconfirmed CR is defined as 1 objective status of CR but not qualifying as a CR or PR, a unconfirmed PR is defined as 1 objective status of PR but not qualifying as CR, PR, or unconfirmed CR. ORR is measured per RECIST 1.1 guidelines.
Time Frame: Up to 5 years post registration or until death
Population: Participants who are eligible and analyzable and had visceral lesions present at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 11
Participants
  Confirmed Complete Response | 0
  Confirmed Partial Response | 0
  Unconfirmed Complete Response | 0
  Unconfirmed Partial Response | 1

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time from date of first registration to date of first documentation of progression or death due to any cause. Patients last known to be alive without report of progression are censored at date of last contact. For a patient to have "progressed", one or more of the following must occur: 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline, as well as an absolute increase of at least 0.5 cm. Unequivocal progression of non-measurable disease in the opinion of the treating physician (an explanation must be provided). Appearance of any new lesion/site. Death due to disease without prior documentation of progression and without symptomatic deterioration.
Time Frame: Up to 5 years post registration or until death
Population: Participants who are eligible and analyzable
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 11 | 27
months | 2.1 [0.7 to 5.5] | 2.3 [1.9 to 6.2]

7. Secondary Outcome: Overall Survival (OS)
Description: Time from date of registration to date of death due to any cause. Participants last known to be alive are censored at date of last contact.
Time Frame: Up to 5 years post registration or until death
Population: Participants who are eligible and analyzable
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 11 | 27
months | 5.2 [1.0 to NA] — Some patients are still alive at the time of reporting so upper confidence boundary is not reportable. | NA [19.1 to NA] — >50% of patients are still alive at the time of reporting so certain data is not reportable.

8. Secondary Outcome: Number of Participants With Gr 1 Through 5 Adverse Events That Are Related to Study Drugs
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported. CTCAE Version 4.0 was used for AE reporting.
Time Frame: Duration of treatment and 5 years follow-up or death, whichever occurs first.
Population: Participants who were eligible and received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab): Cohort B (Non- Visceral): Patients will take up to 4 ml of 1 million PFU/mL T-VEC intralesionally on cycle 1, and up to 4 ml of 100 million PFU/mL T-VEC intralesionally on cycles 2-36, as well as 200 mg of Pembrolizumab taken by IV over 30 minutes on cycles 1-36.
Arm/Group | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab)
Number analyzed (Participants) | 11 | 27
Participants
  Dyspnea | 0 | 1
  Fatigue | 0 | 2
  Hyponatremia | 0 | 1
  Hypoxia | 0 | 1
  Injection site reaction | 0 | 2
  Lymphocyte count decreased | 1 | 0
  Tumor pain | 0 | 1

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 5 years post registration.
Description: CTCAE version 5.0 was used for reporting SAEs and CTCAE version 4.0 was used for reporting toxicities. There were 11 participants in Cohort A and 27 participants in Cohort B that were evaluable for AEs.
Arm/Group | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 1/11 | 0/27
Serious Adverse Events (participants affected / at risk) | 6/11 | 3/27
Other Adverse Events (participants affected / at risk) | 10/11 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) (N=11) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab) (N=27)
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 1
Blurred vision (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Death NOS (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Fever (General disorders) | 1 | 1
Lung infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Visceral): T-VEC + MK-3475 (Pembrolizumab) (N=11) | Cohort B (Non-Visceral): T-VEC + MK-3475 (Pembrolizumab) (N=27)
Anemia (Blood and lymphatic system disorders) | 3 | 8
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 4
Blurred vision (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 0 | 2
Eye disorders-Other (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 4
Bloating (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 5
Diarrhea (Gastrointestinal disorders) | 2 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 11
Proctitis (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 3 | 4
Chills (General disorders) | 3 | 7
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 13
Fever (General disorders) | 2 | 6
Flu like symptoms (General disorders) | 0 | 9
General disorders and admin site conditions - Other (General disorders) | 1 | 1
Injection site reaction (General disorders) | 0 | 6
Malaise (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 2
Pain (General disorders) | 0 | 7
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Anorectal infection (Infections and infestations) | 1 | 0
Infections and infestations-Other (Infections and infestations) | 1 | 1
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 1
Alkaline phosphatase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 2 | 1
Creatinine increased (Investigations) | 1 | 3
Lymphocyte count decreased (Investigations) | 1 | 3
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 1
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 9
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 2 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 5
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 1 | 5
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 4
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Surgical and medical procedures-Other (Surgical and medical procedures) | 0 | 2
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT02965716/Prot_SAP_000.pdf